CLINICAL TRIAL: NCT01797744
Title: Vestibular Rehabilitation for Strokepatients With Dizziness - a Randomized Controlled Trial.
Brief Title: Vestibular Rehabilitation for Strokepatients With Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skåne, Primary health care, Sweden (Unknown)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Associate professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/816
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Stroke; Dizziness
Keywords: Stroke; Dizziness; Vestibular rehabiliation; Balance
MeSH Terms: conditions — Stroke; Dizziness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vestibular rehabiliation (Experimental): Vestibular rehabiliation
  Interventions: Other: Vestibular rehabilitation
- Control group (No Intervention): Usual rehabilitation whitout additional vestibular exercises

INTERVENTIONS:
Other: Vestibular rehabilitation — Usual rehabilitation and four different vestibular rehabilitation exercises, adapted to the individual patient
  Arms: Vestibular rehabiliation

SUMMARY:
Recently, the investigators has shown that dizziness is common among patients with first time stroke and that it affects self perceived health. There are indications that vestibular rehabilitation can have effect of neurological causes of dizziness and vertigo and it therefore seems important to find out if vestibular rehabilitation can affect dizziness among patients with stroke.

The aim of this study is to find out if vestibular rehabilitation can have any effect on function, balance and self-rated health among patients with first time stroke.

ELIGIBILITY:
Inclusion Criteria

• First time stroke with dizziness -

Exclusion Criteria

* Not first time stroke
* No dizziness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The Activities-specific Balance Confidence Scale | Change between baseline and three months after baseline
  Questionnaire. The ABC-scale has proven to be able to identify the influence that vestibular dysfunction can have on daily activities.
EuroQol 5D | Change between baseline and three months after baseline
  Questionnaire. EQ5D consists of a descriptive system comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems, severe problems. The patient indicates his/her state by marking the most appropriate statement. This result in a 1-digit number and the digits for the five dimensions can be combined in a five-digit number, generating 243 possible combinations of response.The EQ5D also consist of the EQ VAS where the patients' record self-rated health on a vertical, visual analogue scale where the individual points can be used as a quantitative measure with zero as worst rated health and 100 as best rated health
The Berg Balance Scale | Change between baseline and three months after baseline
  Balance measures

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Malmo, Sweden

REFERENCES:
- See also: University official website — http://www.med.lu.se